CLINICAL TRIAL: NCT03533348
Title: Preparative Fasting for Contrast-enhanced Computed tomography-a Prospective Randomized Study
Brief Title: Preparative Fasting Before Contrast-enhanced Computed Tomography
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Naiel Bisharat, Head, Department of Medicine D, HaEmek Medical Center, Israel
Other Study IDs: 0167-17-EMC
Record Dates: First submitted 2018-04-30; First posted 2018-05-23 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: X-ray Contrast Media Adverse Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fasting arm: Patients will need at least 4 hours of fasting prior to contrast-enhanced CT scans.
- No fasting: Patients are allowed to eat and drink freely prior to contrast-enhanced CT scans.

SUMMARY:
The study aims to determine whether there is a need for preparative fasting prior to contrast-enhanced computed tomography (CT).

DETAILED DESCRIPTION:
The use of fasting orders for imaging and other procedures is common, this seemingly benign practice can lead to real harms to patients and poor satisfaction with their care. The nothing per os (NPO) order is sometimes used in CT scans because gastrointestinal tract contents can interrupt visualization of the intestinal lumen, but more commonly NPO orders are are thought to protect all supine patients from aspiration during delivery of intravenous contrast. There is limited evidence to support such practice of NPO orders prior to contrast-enhanced CT scans. The authors' main objective is to determine if there is a need for preparative fasting prior to contrast-enhanced CT scans.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing contrast-enhanced CT scans

Exclusion Criteria:

1. Pateints undergoing CT scans while sedated.
2. Patients under the age of 18 years
3. Patients who suffer from a mental disorder that prevents them:

   1. from understanding what s/he consents to and/ or
   2. from choosing decisively and/ or
   3. from communicating his/her consent
4. Patients who were instructed not to eat due to requirements of a specific study (for example.. computed tomography enterography-CTE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are inpatients who are undergoing contrast enhanced computed tomography that will be divided into two cohorts. The first will need at least 4 hours of fasting prior to contrast enhanced computed tomography scans and the second will be allowed to eat and drink freely prior to contrast enhanced computed tomography scans
Sampling Method: Non-Probability Sample
Enrollment: 2148 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Aspiration pneumonitis | Day 1
  Rates of aspiration pneumonitis after contrast-enhanced CT scans

SECONDARY OUTCOMES:
Gastrointestinal symptoms | Hour 1
  Rates of nausea and vomiting after contrast-enhanced CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Naiel Bisharat, MD, Principal Investigator — Emek Medical Center
Locations (1):
- Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Neeman Z, Abu Ata M, Touma E, Saliba W, Barnett-Griness O, Gralnek IM, Rock W, Bisharat N. Is fasting still necessary prior to contrast-enhanced computed tomography? A randomized clinical study. Eur Radiol. 2021 Mar;31(3):1451-1459. doi: 10.1007/s00330-020-07255-0. Epub 2020 Sep 8. PMID 32901302